CLINICAL TRIAL: NCT00143780
Title: Immunogenicity of Pneumococcal Conjugate Vaccine in Adult Allogeneic Bone Marrow Transplant Recipients - Randomized Controlled Trial of Pre-Transplant Donor Immunization
Brief Title: Pneumonia Vaccine in Bone Marrow Transplant Recipients: Usefulness of Donor Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 02-0182-C; P.S.I. Grant No. 02-67
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2005-08

CONDITIONS: Bone Marrow Transplant
Keywords: Bone Marrow Transplant; Pneumonia; Vaccine; Conjugate Vaccine; Polysaccharide Vaccine
MeSH Terms: conditions — Pneumonia

INTERVENTIONS:
Biological: The polysaccharide vaccine used is Pneumovax (Merck vaccines)
Biological: The conjugate vaccine used is Prevnar (Wyeth-Ayerst vaccines)

SUMMARY:
Streptococcus pneumoniae, also known as Pneumococcus, is a common cause of pneumonia in transplant patients. There has been a vaccine available for this infection called Pneumovax. Recently, a new vaccine for this infection called Prevnar has been developed which may be more effective. Vaccinating the bone marrow donor before transplant may boost the recipient's immune response to the vaccine after transplant. This study is done to compare how vaccinating the donor with one of the vaccines will affect the recipient's immune system response to the vaccine.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to assess the immunogenicity of the new pneumococcal conjugate vaccine in a cohort of allogeneic hematopoietic stem cell transplant (allo-HSCT) recipients. This will be done by using an approach of pre-transplant donor immunization with post-transplant recipient immunization. Response will be compared with the standard 23-valent polysaccharide vaccine. It is hypothesized that the conjugate vaccine will provide an enhanced response in this group of immunosuppressed individuals who respond poorly to standard polysaccharide vaccines.

Specific objectives of this study are:

* To determine the antibody response to both vaccines via a measurement of total antibody response and by the opsonophagocytic assay. This assay has the advantage of assessing if patient antibody responses represent truly functional antibodies that display opsonic activity against pneumococcus and is likely better correlated with protective efficacy.
* To determine any acute adverse reactions of the conjugate vaccine in this population. Results of this trial will help lay the foundation for the development of a rationale and optimal pneumococcal vaccination strategy that would prevent significant morbidity in this patient population.

We hypothesize that pneumococcal conjugate vaccine, due to its T-cell dependent response will have greater immunogenicity and protective effect in an allo-HSCT population by using a donor immunization strategy.

ELIGIBILITY:
Inclusion Criteria:

Recipient - Adult male or female marrow recipients who fulfill the following criteria will be eligible for the study: a) Will undergo allogeneic-HSCT in 2-3 weeks.

b) No splenectomy c) Not currently receiving IVIG d) Able to provide written informed consent and comply with study protocol e) Age > 16

Donor - Adult male or female marrow donors who fulfill the following criteria will be eligible for the study:

1. Recipient of donor marrow agrees to participate in study.
2. No prior pneumococcal vaccination within the last 5 years
3. Not on immunosuppressive medication (eg., corticosteroids)
4. No history of immunosuppressive condition that may potentially impair vaccine response eg, systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis
5. No splenectomy
6. Able to provide written informed consent and comply with study protocol
7. Age > 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2002-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of two vaccines via a determination of serotype specific capsular antibody formation and functional antibody formation from donor and recipient serum.

SECONDARY OUTCOMES:
All patients will be called by telephone 24 hours after receiving vaccine to determine if any acute adverse events occurred. Any occurance of pneumococcal disease in recipients for one year post-transplant during the study period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, BSc, MSc, MD, FRCP(C), Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada